CLINICAL TRIAL: NCT05306665
Title: PREventing Pain After Surgery: a Feasibility and Acceptability Study of Acceptance and Commitment Therapy for the Prevention of Chronic Post-surgical Pain (PREPS)
Brief Title: PREventing Pain After Surgery
Acronym: PREPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Samantha Meints, Clinical Psychologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022P002302
Record Dates: First submitted 2022-02-23; First posted 2022-04-01 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Pain, Back; Spinal Stenosis; Disc Herniation; Spondylosis; Spondylolisthesis; Back Injuries
Keywords: Chronic pain; Surgery; opioid; acceptance and commitment therapy; Prevention
MeSH Terms: conditions — Back Pain; Spinal Stenosis; Intervertebral Disc Displacement; Spondylosis; Spondylolisthesis; Back Injuries; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ACT intervention (Experimental): Participants assigned to this arm will complete a 1-day ACT workshop followed by a telephone booster after surgery
  Interventions: Behavioral: ACT intervention
- Treatment As Usual (No Intervention): Participants assigned to this arm will receive treatment as usual.

INTERVENTIONS:
Behavioral: ACT intervention — One day in person workshop + telephone booster
  Arms: ACT intervention

SUMMARY:
The present study aims to adapt and modify a brief presurgical Acceptance and Commitment Therapy (ACT) intervention aimed at preventing the transition to Chronic Post-Surgical Pain (CPSP) and reducing long-term opioid use. Investigators will then assess the acceptability, feasibility, and preliminary efficacy of the finalized intervention to prevent the transition to CPSP and reduce post-surgical opioid use six months following lumbar spine surgery. Finally, investigators will identify psychosocial and psychophysical phenotypes associated with response to this intervention.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo fusion, discectomy, vertebroplasty, kyphoplasty, or foraminotomy
* age 22 and older
* able to communicate fluently in English

Exclusion Criteria:

* inability to complete study procedures due to delirium, dementia, psychosis, or other cognitive impairment
* have a history of severe neurologic movement disorder
* are pregnant or intent to become pregnant during study
* have undergone previous spinal surgery
* have spinal deformity, pseudarthrosis, trauma, infection, or tumor as primary indication for surgery
* have undergone Acceptance and Commitment Therapy in last 2 years

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Helpfulness | Immediately following the ACT workshop
  Treatment Helpfulness Questionnaire (THQ); Item assesses the perceived helpfulness of the ACT workshop and is rated from -5 (extremely harmful) to 5 (extremely helpful).

SECONDARY OUTCOMES:
Pain Interference | 1 month post-op
  Patient Reported Outcomes Measurement Information System-29 (PROMIS-29); Items are rated from 1-5 and then summed with higher scores indicative of greater pain interference
Pain Interference | 3 months post-op
  Patient Reported Outcomes Measurement Information System-29 (PROMIS-29); Items are rated from 1-5 and then summed with higher scores indicative of greater pain interference
Pain Interference | 6 month post-op
  Patient Reported Outcomes Measurement Information System-29 (PROMIS-29); Items are rated from 1-5 and then summed with higher scores indicative of greater pain interference
Treatment Helpfulness | 1 month post-op
  Treatment Helpfulness Questionnaire (THQ); Item assesses the perceived helpfulness of the ACT workshop and is rated from -5 (extremely harmful) to 5 (extremely helpful).
Opioid dose | 1 month post-op
  We will assess daily morphine equivalent doses using the ManageMyPain App and confirm via medical record review
Opioid dose | 3 months post-op
  We will assess daily morphine equivalent doses using the ManageMyPain App and confirm via medical record review
Opioid dose | 6 months post-op
  We will assess daily morphine equivalent doses using the ManageMyPain App and confirm via medical record review
Pain Intensity | 1 month post-op
  Patient Reported Outcomes Measurement Information System-29 (PROMIS-29); Values range from 0-10 with higher scores indicating greater pain intensity
Pain Intensity | 3 months post-op
  Patient Reported Outcomes Measurement Information System-29 (PROMIS-29); Values range from 0-10 with higher scores indicating greater pain intensity
Pain Intensity | 6 months post-op
  Patient Reported Outcomes Measurement Information System-29 (PROMIS-29); Values range from 0-10 with higher scores indicating greater pain intensity
Treatment Credibility | Immediately following ACT workshop
  Credibility and Expectancy Questionnaire (CEQ); 3 items are rated to indicate the logic, success, and confidence in the treatment. Scores are summed with a range from 3-27 where higher scores indicating greater treatment credibility
Treatment Expectancy | Immediately following ACT workshop
  Credibility and Expectancy Questionnaire (CEQ); 3 items are used to assess the likelihood of the success of the therapy to reduce pain and improve function. Scores are summed with a range from 0-29 where higher scores indicate greater expectancy for beneficial treatment outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be stripped of identifiers prior to release for sharing at the time of publication or shortly thereafter. The data will then be made available to approved outside collaborators under a data-sharing agreement that provides for (1) commitment to using the data only for research purposes; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying the data after analyses are completed. Further, the data will be shared via publication and/or public presentations.
Supporting Information: Study Protocol
Time Frame: The time of publication or shortly afterward.